CLINICAL TRIAL: NCT04841954
Title: Hemp Seed Awareness
Acronym: ARCHANGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 49RC21_0048
Record Dates: First submitted 2021-04-02; First posted 2021-04-12 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prick-test (Experimental)
  Interventions: Diagnostic Test: hemp prick-test

INTERVENTIONS:
Diagnostic Test: hemp prick-test — hemp seed and flower prick-test

SUMMARY:
Hemp is a plant of the Cannabaceae family. Cannabis sativa, derived from female flowers, is the first illicit substance used by adolescents and is a major public health problem. Its psycho-active effects come from tetrahydrocannabinol (THC).

Unlike recreational cannabis, industrial hemp derived from cannabis sativa has a high level of cannabidiol (CBD) but a negligible level of tetrahydrocannabinol. Its seeds are now consumed in various forms and generate increasing interest. Seeds have many nutritional benefits.

It seems important to take an interest in hemp, given the recent expansion of medical cannabis and the increasing use of cannabis for recreational purposes. It is incriminated in various allergies (contact dermatitis, asthma, rhinoconjunctivitis) but also in the occurrence of anaphylaxis to certain foods by cross-allergy in atopic subjects, in association with an Lipid-Transfer Proteins (LTP protein), present in the flower of Cannabis sativa.

Unlike the allergy to recreational cannabis, the allergenicity of hemp seeds is little studied.

Hemp seed can cause severe anaphylactic reactions. In all reported cases, the prick-tests were positive for the seeds. Often, patients had never been in contact with hemp seeds but had already been exposed to cannabis by respiratory or manual routes.

The investigators hypothesize that sensitization by the skin or respiratory route (cannabis smokers, passive exposure to cannabis, workers exposed to hemp, etc.) could lead to the development of a food allergy to hemp seed.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Patient referred to the Allergology Unit of the Hospital of Angers, in consultation or in Hospitalization - for conducting prick-tests
* Patient affiliated or beneficiary of a social security scheme
* Patient with informed consent

Exclusion Criteria:

* Pregnant women, parturients
* Persons deprived of liberty by administrative or judicial decision
* Persons receiving psychiatric care under duress
* Adults under legal protection measure
* People out of state to express consent
* people not able to understand French language
* Patients whose skin reactivity prevents interpretation of tests (patients who cannot interrupt anti-histamines or have severe eczema)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Positive prick-test | Day 1
  To assess the prevalence of hemp seed sensitization in the allergy consulting population

SECONDARY OUTCOMES:
history of hemp use | Day 1
  To study the association between sensitization to hemp seed and patient characteristics

CONTACTS AND LOCATIONS:
Locations (1):
- MORISSET Martine, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided